CLINICAL TRIAL: NCT00468247
Title: A Prospective,Open,Multicentre,RCT to Assess the Safety & Efficacy of Navigator v Conventional Care in Post-op Cardiac Surgery Patients Undergoing CABG &/or Heart Valve Repair/Replacement Utilising Heart Lung Perfusion Pump(The NAV-1 Study)
Brief Title: Registration Enabling Study of the Safety and Efficacy of the Use of the Navigator Circulatory Management System
Acronym: NAV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Applied Physiology Pty Ltd (Other)
Collaborators: Trident Clinical Research Pty Ltd (Industry)
Responsible Party: Vickie Edwards, Applied Physiology Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP2006-01
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Critical Illness; Intensive Care
Keywords: mean systemic pressure; fluid therapy; closed loop control; circulation modelling
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Device , Navigator used for guiding haemodynamic care
  Interventions: Device: Navigator
- 2 (Placebo Comparator): Conventional care
  Interventions: Other: Conventional care

INTERVENTIONS:
Device: Navigator — Navigator circulatory mgt system
  Arms: 1
Other: Conventional care — Conventional haemodynamic care
  Arms: 2

SUMMARY:
A multicentre, open, RCT to assess the safety and efficacy of the Navigator Guided Circulatory Management System versus conventional care in post-operative cardiac surgery patients. The purpose of the study is to demonstrate that the real time acquisition and subsequent processing and display of data produced by the Navigator guided circulatory management system provides the clinician with appropriate data and guidance to achieve and maintain a prescribed target haemodynamic stability in the post operative patient when compared to conventional care in an Intensive Care Unit setting.

DETAILED DESCRIPTION:
Protocol No. AP2006-01

Study title: A Prospective, Open, Randomised, Multicentre, Controlled Group Study to Assess the Safety and Efficacy of Navigator versus Conventional Care in Postoperative Cardiac Surgery Patients Undergoing Coronary Bypass Grafting and or Heart Valve Repair or Replacement Utilizing Heart Lung Perfusion Pump.

Acronym: NAV 1

Type of study: Device Trial

Sponsor: Applied Physiology Pty Ltd

Study device: Navigator Guided Circulatory Care Management System

Route of Administration: Via Touch Panel Computer, externally connected to the bedside physiological monitor in a critical care environment

Study centres: Six Australian centres

Study design: Multicentre, open, randomised, controlled group study

Total sample size: One hundred completed patients, 50 in each arm

Study population: Post operative coronary bypass and heart valve repair or replacement patients admitted to a Cardiac Intensive Care or Intensive Care Unit. Surgery must involve the use of a heart lung perfusion pump and the patient must have a functioning arterial line and Swan Ganz catheter in situ to enable the measurement of Cardiac Output, Mean Arterial Pressure, and Right Atrial Pressure.

Study regimen: Following surgery, and after meeting inclusion and exclusion criteria, patients will be randomised on admission to ICU to receive care guided by Navigator or conventional care during their ICU stay while CO is being monitored. All patients will be connected to the Navigator; the screen of the patients in the control group will have the graphical section blank, the right hand side will display actual values of MAP, CO and RAP as slaved from the bedside monitor, along with the patient's screening and randomisation number and initials. The arm of the study to which the patient has been randomised ;control/Navigator, will also be shown.

Endpoints:

Primary: The primary efficacy endpoint is the average distance to the central point of the target cardiovascular zone over the period the patient is connected to Navigator.

Secondary: Secondary endpoints for the trial will be:

* Percentage time in the target cardiovascular zone over the period the patient is connected to the Navigator
* Clinically significant atrial fibrillation over the period the patient is connected to the Navigator. This is defined as irregular supraventricular rhythm with an absence of discrete P waves lasting more than ten minutes documented and confirmed with an ECG
* Multiple organ function, as assessed using the SOFA score, calculated daily
* Navigator device related adverse events and device failures

Statistical analysis: The primary and secondary endpoints and all safety data will be analysed on the randomised Intention-to-treat population.The ITT population will include all individuals who are randomised. The analysis will compare the primary efficacy endpoint between the two randomised treatment groups using independent t tests. The secondary analyses will compare the secondary endpoints between the two randomised treatment groups using independent t-tests, Chi-square tests and Fisher's exact tests as appropriate.

Study Period: From the first pre-surgery screening visit to the post operative follow up visit, approximately six weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older
2. Undergoing elective cardiac surgery where surgery involves the use of a heart-lung perfusion pump
3. Will have an arterial line and Swan Ganz catheter in situ
4. Require invasive measurement of Cardiac Output (CO), Mean Arterial Pressure (MAP) and Right Atrial Pressure (RAP)
5. Are able and willing to provide written informed consent to participate in the study

Exclusion Criteria:

1. Women who are lactating or pregnant
2. Require Extracorporeal Membrane Oxygenation
3. Present at baseline screening or immediately prior to randomisation in the ICU with atrial fibrillation (irregular supraventricular rhythm, not due to ectopic complexes with an absence of discrete P-waves lasting more than 10 minutes documented and confirmed with an ECG)
4. Intra-operative surgical treatment for atrial fibrillation
5. Surgery for left atrial reduction
6. Patients with left ventricular assist devices
7. Patients with permanent pacemakers in situ
8. Deemed by the investigator to be uncooperative or unsuitable for inclusion into this trial
9. Have a medical condition that in the opinion of the investigator would jeopardise the patient's safety by participating in this trial
10. Current participation in another drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Average distance to central point of the target cardiovascular zone while connected to the device | Time connected to Navigator device

SECONDARY OUTCOMES:
Percentage time in the target cardiovascular zone while connected to device | Time connected to Navigator device
Clinically significant AF while connected to device | Time connected to Navigator device
Multiple organ function (SOFA score) | From connection to Navigator device to hospital discharge
Device-related adverse events and device failures | Time connected to Navigator device

CONTACTS AND LOCATIONS:
Overall Officials: Yugan Mudaliar, PhD, Principal Investigator — Western Sydney Area Health Service; Geoff Parkin, PhD, Study Director — Monash Medical Centre
Locations (7):
- Australia (7):
  - St Vincent's Public Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Private Hospital, Sydney, New South Wales
  - Westmead Public Hospital, Sydney, New South Wales
  - St George Public Hospital, Sydney, New South Wales
  - Monash Medical Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria

REFERENCES:
- [Background] Parkin WG. Volume state control - a new approach. Crit Care Resusc. 1999 Sep;1(3):311-21. PMID 16603021
- [Derived] Pellegrino VA, Mudaliar Y, Gopalakrishnan M, Horton MD, Killick CJ, Parkin WG, Playford HR, Raper RF. Computer based haemodynamic guidance system is effective and safe in management of postoperative cardiac surgery patients. Anaesth Intensive Care. 2011 Mar;39(2):191-201. doi: 10.1177/0310057X1103900207. PMID 21485666
- See also: Related Info — http://www.applied-physiology.com